CLINICAL TRIAL: NCT05575544
Title: A Randomized Control Trial to Determine Whether Electroacupuncture(EA) Intervention With Morphine Can Reduce the Intraoperative Pain and Early Post-operative Complications in Patients Undergoing Catheter Ablation of Atrial Fibrillation.
Brief Title: Electroacupuncture Intervention in Catheter Ablation of Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, deputy director of cardiology department of Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EAAF
Record Dates: First submitted 2022-09-23; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Acupuncture Therapy; Morphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left PVI ablation electroacupuncture group (Experimental): Patient undergo right pulmonary vein isolation under general anesthesia.After successful isolation of the right pulmonary vein, use a 25-gauge stainless steel millineedle of different lengths to be ordered sequentially according to the acupuncture point prescription.Acupuncture was performed at Hegu and Neiguan points on the left side of the patient.After the manual acupuncture, the point was continuously stimulated by an electrical stimulator to analgesia,the frequency is 200 times / min, the pulse frequency is 3 ~ 4Hz. The output intensity is subject to the patient's tolerance, generally 20mA.The electroneedle stimulates until the end of the left pulmonary vein isolation.
  Interventions: Procedure: Acupuncture plus morphine
- Right PVI ablation electroacupuncture group (Experimental): Patient undergo left pulmonary vein isolation under general anesthesia.After successful isolation of the left pulmonary vein, use a 25-gauge stainless steel millineedle of different lengths to be ordered sequentially according to the acupuncture point prescription.Acupuncture was performed at Hegu and Neiguan points on the left side of the patient.After the manual acupuncture, the point was continuously stimulated by an electrical stimulator to analgesia,the frequency is 200 times / min, the pulse frequency is 3 ~ 4Hz. The output intensity is subject to the patient's tolerance, generally 20mA.The electroneedle stimulates until the end of the right pulmonary vein isolation.
  Interventions: Procedure: Acupuncture plus morphine

INTERVENTIONS:
Procedure: Acupuncture plus morphine — The acupuncture was combined with intravenous use of morphine to achieve anesthesia during the ablation procedure

SUMMARY:
This is a randomized control trial to determine whether electroacupuncture(EA) intervention with Morphine can reduce the intraoperative pain and early post-operative complications in patients undergoing catheter ablation of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old;
2. Atrial fibrillation
3. Nonresponse or intolerance to ≥1 antiarrhythmic drug.

Exclusion Criteria:

1. A history of allergy to acupuncture;
2. With uncontrolled congestive heart failure;
3. Having significant valvular disease;
4. Having moderate-to-severe pulmonary hypertension;
5. With myocardial infarction or stroke within 6 months of screening;
6. With Significant congenital heart disease;
7. Ejection fraction was <40% measured by echocardiography;
8. Allergic to contrast media;
9. Contraindication to anticoagulation medications;
10. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD);
11. Left atrial thrombus;
12. Having any contraindication to right or left sided heart catheterization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-11 (Estimated); Primary Completion 2023-10-11 (Estimated); Study Completion 2023-10-13 (Estimated)

PRIMARY OUTCOMES:
The severity of intraprocedural pain during the catheter ablation procedure | up to 1 month after enrollment
  Pain was assessed by Visual Analogue Score (VAS).VAS is one of the commonly used pain scoring standards. The full name is the visual simulation scoring method. The pain is divided into 10 points, 2 points for no pain, 10 points for severe pain, and the middle part for different degrees of pain.To compare the scores of patients during pulmonary vein isolation procedure.
The severity of intraprocedural nausea during the catheter ablation procedure | up to 1 month after enrollment
  The incidence of nausea, vomiting and retching within 12 hours after operation was recorded, including 3 dimensions of symptom experience time, frequency and severity, with 8 items in total. 0~4 points shall be used for 5 grades. 0 points means none at all, and 4 points means very serious and intolerable.

SECONDARY OUTCOMES:
The dose of morphine used during the catheter ablation procedure | up to 1 month after enrollment
  To compare the dose of morphine used during pulmonary vein isolation procedure.
the change of blood pressure during the catheter ablation procedure | up to 1 months after enrollment
  Record the changes of blood pressure during the catheter ablation procedure
Change of the the radio of IL6/IL10 before and after the ablation procedure | up to 1 months after enrollment
Incidence of complications | up to 6 months after enrollment
  death, atrio-esophageal fistula, cardiac tamponade/perforation, myocardial infarction, stroke/cerebrovascular accident, thromboembolism, diaphragmatic paralysis, pneumothorax, pleural effusion, heart block, pulmonary vein stenosis, pulmonary edema, left atrial thrombus, pericarditis and major vascular access complication or bleeding